**Grant Title:** The emergence of abstract structure knowledge across learning and sleep

NCT number: NCT05746299

**Date:** June 17, 2025

## **Statistical Analysis Plan**

For Aim 1, the outcome measure is accuracy (0-100%) on the missing feature task for the Modular category in Stage 2. The statistical method we will use to assess this outcome measure will be a two-sample t-test to compare accuracy on the new Modular category in Stage 2 across groups (Congruent vs. Incongruent).

For Aim 2, the outcome measure is accuracy (0-100%) on the missing feature task for the Modular category in Stage 2. The statistical method we will use to assess this outcome measure will be a two-sample t-test to compare accuracy across groups (Congruent vs. Incongruent, Awake vs. Sleep).

Our statistical methods are appropriate given comparable research on category learning and structure learning.